CLINICAL TRIAL: NCT06171516
Title: Internet-based Cognitive Behavioral Therapy for Individuals With Gambling Disorder in Indonesia: a Pilot and Feasibility Study
Brief Title: Internet-based Cognitive Behavioral Therapy for Individuals With Gambling Disorder in Indonesia
Acronym: ICBT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Flinders University (Other)
Responsible Party: Principal Investigator, Kristiana Siste, Dr. dr. Kristiana Siste, SpKJ(K) - Head of Department of Psychiatry, Faculty of Medicine, Indonesia University, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KET-992-2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based Cognitive Behavioral Therapy (Experimental): 10 guided therapy sessions (once-weekly) with each session lasting 20 minutes.
  Interventions: Behavioral: iCBT

INTERVENTIONS:
Behavioral: iCBT — All participants will undergo 10 guided therapy sessions (once-weekly) with each session lasting 20 minutes. The therapy module will be given as an online self-learning source via videos in a website specifically developed for this training. The videos will divide the module content into several parts with each video lasting about 10 minutes.

SUMMARY:
Gambling disorder (GD) has become a wide concern in Indonesia, as many negative consequences aroused from this psychiatric condition. Prompt treatment with appropriate method of delivery is required to achieve optimal outcome in GD patients. This study aims to determine the effectiveness and feasibility of internet-based cognitive behavioral therapy (iCBT) in treating GD.

This non-randomised pilot and feasibility study will recruit 20 people with GD. All participants will receive the iCBT intervention through self-learning videos and guided weekly group sessions. The effectiveness of the intervention will be assessed at baseline (week 0), post-treatment completion (week 10), and 6 weeks post-treatment (week 16).

Expanded access of the iCBT module will not be available until after the study completion.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18-59 years old;
* be screened as probable pathological gambler based on South Oaks Gambling Screen (SOGS);
* have access to electronic devices (ie, smartphone, mobile tablet, personal computer) with internet connection;
* be proficient in Indonesian language;
* have agreed to take part in the study by filling out the informed consent form.

Exclusion Criteria:

* have severe mental disorders or intellectual disabilities;
* have extreme agitation that hinder instrument fill out and adequate cognitive behavior therapy participation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Gambling symptom severity | G-SAS will be assessed at baseline (week 0), post-treatment (week 6), and follow-up (week 16)
  a decrease in Gambling Symptom Assessment Scale (G-SAS) score
Problem gambling severity | PGSI will be assessed at baseline (week 0), post-treatment (week 6), and follow-up (week 16)
  a decrease in Problem Gambling Severity Index score
Gambling urges | GUS will be assessed at baseline (week 0), post-treatment (week 6), and follow-up (week 16)
  a decrease in Gambling Urge Scale (GUS) score
Gambling-related cognitive distortions | GRCS will be assessed at baseline (week 0), post-treatment (week 6), and follow-up (week 16)
  a decrease in Gambling Related Cognitions Scale (GRCS) score

SECONDARY OUTCOMES:
Nonspecific psychological distress | SRQ-20 will be assessed at baseline (week 0), post-treatment (week 6), and follow-up (week 16)
  a decrease in Self Rating Questionnaire-20 (SRQ-20) score
Subjective quality of life | WHOQOL-BREF will be assessed at baseline (week 0), post-treatment (week 6), and follow-up (week 16)
  an increase in World Health Organization Quality-of-Life Scale (WHOQOL-BREF) score